CLINICAL TRIAL: NCT03502551
Title: ED Treatment of Suicidal Patients With Ketamine Infusion
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial never received funding.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1197884
Record Dates: First submitted 2018-03-01; First posted 2018-04-18 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Suicide; Suicidal Ideation
Keywords: ketamine; suicide
MeSH Terms: conditions — Suicide; Suicidal Ideation | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with Ketamine (Experimental): In this arm an IV infusion of 0.5 mg/kg of ketamine will be administered over 40 minutes.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine infusion (0.5 mg/kg) over 40 minutes.
  Other Names: Ketalar

SUMMARY:
This study aims to determine if a single intravenous (IV) dose of ketamine given in the emergency department (ED) can provide a long term reduction in suicidal ideation, lower time to ED discharge, and increase discharge to home or voluntary treatment facilities all while being safe.

DETAILED DESCRIPTION:
Suicide has risen to the 2nd leading cause of death in Americans aged 10 to 34, and is the10th leading cause of death overall. Globally, the World Health Organization estimates one person dies of suicide every 40 seconds. Despite its lethality, no recognized acute treatments for suicidality exist. Recently, ketamine, an N-methyl-D-aspartate (NMDA) receptor agonist, has been shown to rapidly reduce suicidality in small studies in psychiatric settings. However, most patients with acute suicidal thoughts are treated initially in Emergency Departments (EDs). Delays in treatment have both short and long term impacts on recovery as patients spend longer time frames in an actively suicidal state.

Identifying a rapid and effective treatment for suicidal ideation that can be administered in the ED would have a profound impact on the emergent management of patients with suicidal thoughts. Ketamine is an FDA approved medication that is commonly used in EDs for multiple indications. EDs have the familiarity, facilities and personnel to safely administer IV ketamine.

Ketamine is regularly used in EDs in high doses for procedural sedation in adults and children. It is also used in high doses as a sedative for acutely agitated patients. In low-doses ketamine is frequently used for its analgesic properties and is considered safe.

Ketamine has also been safely used in the pre-hospital setting. In a recent joint policy statement of the American College of Emergency Physicians recommended the use of low-dose ketamine for pain in control with a safety profile comparable to other intravenous analgesia such as morphine.

Use of Ketamine to rapidly reduce suicidality may facilitate a safe and faster transition of acutely suicidal patients to outpatient treatment. Such treatment potentially shortens these patients' ED and hospital lengths of stay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Chief complaint of suicidal thoughts with a MADRS-SI score > 3
* Major depressive episode with MADRS > 19 (moderate to severe)

Exclusion Criteria:

* Pregnancy
* Psychosis
* Acute intoxication with alcohol or illicit drugs
* Acute withdrawal from alcohol or illicit drugs
* Adults otherwise unable to consent
* Concurrent, active medical illness requiring medical hospitalization
* Inability to follow-up including no permanent address or valid telephone number
* Patients unable to attend outpatient follow-up (no medical insurance, refusal to follow-up, no established care provider)
* Specific contraindication to the use of ketamine (concern for increased intracranial or intraocular pressure, known allergy to ketamine)
* Greater than 12 hours from time of ED presentation
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation at 24 hours post-infusion | 24 hours post-infusion
  Suicidal ideation as measured by the Montgomery-Asberg Depression Scale (MARDS) will be assessed at 24 hours post-infusion of ketamine. The scale is a series of 10 questions each having a possible score of 0-6. Total scores are reported on a scale from 0-60, with lower numbers indicating less depression and higher numbers indicative of increasing depression.
Incidence of Discharge to Outpatient vs. Inpatient Facilities | Through ED stay, an average of 53 hours
  The investigators will collect information about what location patients enrolled in this study are discharged to (E.g. home, outpatient crisis residential facility, inpatient psychiatric hospital, admission to general hospital).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 week from enrollment.
  Patients will be monitored for adverse events during the course of this study.

SECONDARY OUTCOMES:
Overall MARDS score | 1 hour, 3 days, and 1 week post-infusion
  The MARDS will be administered regularly throughout the study and will serve as a measure of suicidal ideation. The scale is a series of 10 questions each having a possible score of 0-6. Total scores are reported on a scale from 0-60, with lower numbers indicating less depression and higher numbers indicative of increasing depression.
MARDS Suicidal Ideation (MARDS-SI) score | 1 hour, 3 days, and 1 week post-infusion
  The MARDS will be administered regularly throughout the study and will serve as a measure of suicidal ideation. Item 10 on the MARDS serves to specifically measure suicidal ideation with a score of 4 or greater being considered to indicate marked suicidal ideations.
Scale for Suicide Ideation-5 (SSI5) score | 1 hour, 3 days, and 1 week post-infusion
  The Scale for Suicide Ideation (SSI) will be administered regularly throughout the study and will serve as a measure of suicidal ideation. Items 1-5 on the SSI serves to specifically measure suicidal ideation. Each of the five questions on the scale have three possible answers with scores ranging from 0 (no suicidal ideation) to 2 (increased suicidal ideation). To compute the SSI5, the scores from each of the five questions are added together to give an overall score from 0-10, where 0 is no suicidal ideation and 10 is increased suicidal ideation.
ED length of stay | Through ED stay, an average of 53 hours
  The investigators will measure the amount of time that patients in this study remain in the ED before being discharged or transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Moulin, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price RB, Iosifescu DV, Murrough JW, Chang LC, Al Jurdi RK, Iqbal SZ, Soleimani L, Charney DS, Foulkes AL, Mathew SJ. Effects of ketamine on explicit and implicit suicidal cognition: a randomized controlled trial in treatment-resistant depression. Depress Anxiety. 2014 Apr;31(4):335-43. doi: 10.1002/da.22253. Epub 2014 Mar 25. PMID 24668760
- [Background] Zarate CA Jr, Brutsche NE, Ibrahim L, Franco-Chaves J, Diazgranados N, Cravchik A, Selter J, Marquardt CA, Liberty V, Luckenbaugh DA. Replication of ketamine's antidepressant efficacy in bipolar depression: a randomized controlled add-on trial. Biol Psychiatry. 2012 Jun 1;71(11):939-46. doi: 10.1016/j.biopsych.2011.12.010. Epub 2012 Jan 31. PMID 22297150
- [Background] DiazGranados N, Ibrahim LA, Brutsche NE, Ameli R, Henter ID, Luckenbaugh DA, Machado-Vieira R, Zarate CA Jr. Rapid resolution of suicidal ideation after a single infusion of an N-methyl-D-aspartate antagonist in patients with treatment-resistant major depressive disorder. J Clin Psychiatry. 2010 Dec;71(12):1605-11. doi: 10.4088/JCP.09m05327blu. Epub 2010 Jul 13. PMID 20673547
- [Background] Murrough JW, Soleimani L, DeWilde KE, Collins KA, Lapidus KA, Iacoviello BM, Lener M, Kautz M, Kim J, Stern JB, Price RB, Perez AM, Brallier JW, Rodriguez GJ, Goodman WK, Iosifescu DV, Charney DS. Ketamine for rapid reduction of suicidal ideation: a randomized controlled trial. Psychol Med. 2015 Dec;45(16):3571-80. doi: 10.1017/S0033291715001506. Epub 2015 Aug 12. PMID 26266877
- [Background] Zhu JM, Singhal A, Hsia RY. Emergency Department Length-Of-Stay For Psychiatric Visits Was Significantly Longer Than For Nonpsychiatric Visits, 2002-11. Health Aff (Millwood). 2016 Sep 1;35(9):1698-706. doi: 10.1377/hlthaff.2016.0344. PMID 27605653
- [Background] Godwin SA, Burton JH, Gerardo CJ, Hatten BW, Mace SE, Silvers SM, Fesmire FM; American College of Emergency Physicians. Clinical policy: procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2014 Feb;63(2):247-58.e18. doi: 10.1016/j.annemergmed.2013.10.015. PMID 24438649
- [Background] Hopper AB, Vilke GM, Castillo EM, Campillo A, Davie T, Wilson MP. Ketamine use for acute agitation in the emergency department. J Emerg Med. 2015 Jun;48(6):712-9. doi: 10.1016/j.jemermed.2015.02.019. Epub 2015 Apr 2. PMID 25843924
- [Background] Miner JR, Moore JC, Austad EJ, Plummer D, Hubbard L, Gray RO. Randomized, double-blinded, clinical trial of propofol, 1:1 propofol/ketamine, and 4:1 propofol/ketamine for deep procedural sedation in the emergency department. Ann Emerg Med. 2015 May;65(5):479-488.e2. doi: 10.1016/j.annemergmed.2014.08.046. Epub 2014 Oct 16. PMID 25441247
- [Background] Patanwala AE, McKinney CB, Erstad BL, Sakles JC. Retrospective analysis of etomidate versus ketamine for first-pass intubation success in an academic emergency department. Acad Emerg Med. 2014 Jan;21(1):87-91. doi: 10.1111/acem.12292. PMID 24552528
- [Background] Sin B, Ternas T, Motov SM. The use of subdissociative-dose ketamine for acute pain in the emergency department. Acad Emerg Med. 2015 Mar;22(3):251-7. doi: 10.1111/acem.12604. Epub 2015 Feb 25. PMID 25716117
- [Background] Grossimlinghaus I, Falkai P, Gaebel W, Hasan A, Janner M, Janssen B, Reich-Erkelenz D, Gruber L, Bottcher V, Wobrock T, Zielasek J; LVR-Klinikverbund. [Assessment of quality indicators with routine data: Presentation of a feasibility test in ten specialist clinics for psychiatry and psychotherapy]. Nervenarzt. 2015 Nov;86(11):1393-9. doi: 10.1007/s00115-015-4357-y. German. PMID 26122639
- [Background] American College of Emergency Physicians Clinical Policies Subcommittee (Writing Committee) on the Adult Psychiatric Patient; Nazarian DJ, Broder JS, Thiessen MEW, Wilson MP, Zun LS, Brown MD. Clinical Policy: Critical Issues in the Diagnosis and Management of the Adult Psychiatric Patient in the Emergency Department. Ann Emerg Med. 2017 Apr;69(4):480-498. doi: 10.1016/j.annemergmed.2017.01.036. No abstract available. PMID 28335913
- [Background] Pourmand A, Mazer-Amirshahi M, Royall C, Alhawas R, Shesser R. Low dose ketamine use in the emergency department, a new direction in pain management. Am J Emerg Med. 2017 Jun;35(6):918-921. doi: 10.1016/j.ajem.2017.03.005. Epub 2017 Mar 2. PMID 28285863
- [Background] Lee EN, Lee JH. The Effects of Low-Dose Ketamine on Acute Pain in an Emergency Setting: A Systematic Review and Meta-Analysis. PLoS One. 2016 Oct 27;11(10):e0165461. doi: 10.1371/journal.pone.0165461. eCollection 2016. PMID 27788221
- [Background] Scaggs TR, Glass DM, Hutchcraft MG, Weir WB. Prehospital Ketamine is a Safe and Effective Treatment for Excited Delirium in a Community Hospital Based EMS System. Prehosp Disaster Med. 2016 Oct;31(5):563-9. doi: 10.1017/S1049023X16000662. Epub 2016 Aug 12. PMID 27517801
- [Background] Jennings PA, Cameron P, Bernard S. Ketamine as an analgesic in the pre-hospital setting: a systematic review. Acta Anaesthesiol Scand. 2011 Jul;55(6):638-43. doi: 10.1111/j.1399-6576.2011.02446.x. Epub 2011 May 16. PMID 21574967
- [Background] Ballard ED, Luckenbaugh DA, Richards EM, Walls TL, Brutsche NE, Ameli R, Niciu MJ, Vande Voort JL, Zarate CA Jr. Assessing measures of suicidal ideation in clinical trials with a rapid-acting antidepressant. J Psychiatr Res. 2015 Sep;68:68-73. doi: 10.1016/j.jpsychires.2015.06.003. Epub 2015 Jun 16. PMID 26228403
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082
- [Background] McGirr A, Berlim MT, Bond DJ, Fleck MP, Yatham LN, Lam RW. A systematic review and meta-analysis of randomized, double-blind, placebo-controlled trials of ketamine in the rapid treatment of major depressive episodes. Psychol Med. 2015 Mar;45(4):693-704. doi: 10.1017/S0033291714001603. Epub 2014 Jul 10. PMID 25010396